CLINICAL TRIAL: NCT05116800
Title: A Phase 2 Study of 9-ING-41, a Glycogen Synthase Kinase-3 Beta (GSK-3β) Inhibitor, Combined With Chemotherapy in Advanced Soft Tissue and Bone Sarcomas
Brief Title: Phase 2 Study of 9-ING-41 With Chemotherapy in Sarcoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: IND withdrawn
Sponsor: Brown University (Other)
Collaborators: Actuate Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Br 398
Record Dates: First submitted 2021-11-02; First posted 2021-11-11 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Soft Tissue Sarcoma; Undifferentiated Pleomorphic Sarcoma; Myxofibrosarcoma; Leiomyosarcoma; Liposarcoma; Angiosarcoma; Synovial Sarcoma; Rhabdomyosarcoma; Spindle Cell Sarcoma; High Grade Sarcoma; Bone Sarcoma; Osteosarcoma; Ewing Sarcoma of Bone
MeSH Terms: conditions — Sarcoma; Histiocytoma, Malignant Fibrous; Dermatofibrosarcoma; Leiomyosarcoma; Liposarcoma; Hemangiosarcoma; Sarcoma, Synovial; Rhabdomyosarcoma; Bone Neoplasms; Osteosarcoma | interventions — Gemcitabine; 3-(5-fluorobenzofuran-3-yl)-4-(5-methyl-5H-(1,3)dioxolo(4,5-f)indol-7-yl)-pyrrole-2,5-dione; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stratum A: Soft Tissue Sarcoma (Experimental): Patients with advanced soft tissue sarcoma previously treated with 0-3 prior lines of systemic therapy will receive 9-ING-41 twice weekly with gemcitabine on days 1 and 8 and docetaxel on day 8 of a 21-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine; Drug: 9-ING-41; Drug: Docetaxel
- Stratum B: Bone Sarcoma (Experimental): Patients with relapsed or refractory bone sarcoma previously treated with at least one line of systemic therapy will receive 9-ING-41 twice weekly with gemcitabine on days 1 and 8 and docetaxel on day 8 of a 21-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine; Drug: 9-ING-41; Drug: Docetaxel

INTERVENTIONS:
Drug: Gemcitabine — Patients will receive 9.3 mg/kg 9-ING-41 twice weekly with 900 mg/m2 gemcitabine on days 1 and 8 and 75 mg/m2 docetaxel on day 8 of a 21-day cycle until disease progression or unacceptable toxicity.
Drug: 9-ING-41 — Patients will receive 9.3 mg/kg 9-ING-41 twice weekly with 900 mg/m2 gemcitabine on days 1 and 8 and 75 mg/m2 docetaxel on day 8 of a 21-day cycle until disease progression or unacceptable toxicity.
Drug: Docetaxel — Patients will receive 9.3 mg/kg 9-ING-41 twice weekly with 900 mg/m2 gemcitabine on days 1 and 8 and 75 mg/m2 docetaxel on day 8 of a 21-day cycle until disease progression or unacceptable toxicity.

SUMMARY:
This is an open label, two-stratum, phase 2 clinical trial evaluating the efficacy of 9-ING-41 in combination with gemcitabine/docetaxel in patients ≥10 years of age with advanced sarcoma. 9-ING-41 in combination with gemcitabine and docetaxel will lead to sustained disease control and/or increase the rates of objective response in patients with unresectable or metastatic soft tissue and bone sarcomas.

ELIGIBILITY:
Inclusion Criteria:

* Stratum A: Patients must have histologically confirmed grade 2 or 3 soft tissue sarcoma that is locally advanced and unresectable, or metastatic, consisting of one of the following subtypes: undifferentiated pleomorphic sarcoma (malignant fibrous histiocytoma), myxofibrosarcoma, leiomyosarcoma, liposarcoma (excluding well-differentiated), angiosarcoma, synovial sarcoma, rhabdomyosarcoma, spindle cell sarcoma and high-grade sarcoma NOS.
* Stratum B: Patients must have histologically confirmed bone sarcoma that is relapsed or refractory following front-line therapy consisting of one of the following subtypes: osteosarcoma and Ewing sarcoma.
* Patients must have at least one site of measurable disease by RECIST 1.1. See Section 12 (Measurement of Effect) for the evaluation of measurable disease.
* Stratum A: No more than three prior lines of systemic therapy. Of note, anthracycline-based chemotherapy is generally considered first-line therapy. Previously untreated patients may be enrolled at the discretion of the treating investigator.
* Stratum B: At least one prior line of systemic therapy.
* Age ≥10 years.
* Lansky score ≥50 for patients <16 years or ECOG performance status ≤2 for patients ≥16 years (Karnofsky ≥50%, see Appendix A).
* Life expectancy of greater than 12 weeks.
* Patients must have adequate organ and marrow function as defined below:

  * Hemoglobin ≥8 g/dl
  * absolute neutrophil count ≥1,000/mcL
  * platelets ≥100,000/mcL (transfusion independent)
  * total bilirubin ≤1.5x institutional upper limit of normal (ULN) (<3.0 mg/dL and direct bilirubin <1.5 mg/dL if documented Gilbert's syndrome)
  * AST(SGOT)/ALT(SGPT) ≤2.5x institutional ULN (≤ 5 x ULN if liver metastases present)
  * creatinine ≤1.5x institutional ULN OR
  * glomerular filtration rate (GFR) ≥50 mL/min/1.73 m2
  * PT/INR ≤1.5x institutional ULN
  * Amylase and lipase ≤1.5x institutional ULN
* Washout period prior to Cycle 1, Day 1:

  * ≥ 21 days since last dose of chemotherapy, immunotherapy, or therapeutic radiation treatment.
  * ≥ 28 days since last tyrosine kinase inhibitor (or 5 half-lives, whichever is shorter).
  * ≥ 7 days since last focal palliative radiation treatment.
  * ≥ 28 days since major surgical procedure.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Women of child-bearing potential must have a negative serum or urine pregnancy test at registration and within 7 days of first study therapy.
* The effects of 9-ING-41 on the developing human fetus are unknown. For this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women may not be breastfeeding during study participation. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 90 days after completion of 9-ING-41 administration.
* Patients must agree to provide tumor tissue, either fresh or archival specimen of primary tumor and/or metastatic lesion. If tumor tissue is not available, then discuss with principal investigator.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with sarcoma histologies other than those listed above will be excluded.
* Prior treatment with 9-ING-41, gemcitabine, or docetaxel.
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
* Patients who are receiving any other investigational agents for treatment of their sarcoma.
* Patients who are pregnant or lactating.
* Patients with untreated brain or meningeal metastases. Subjects with history of metastases are eligible provided they do not require ongoing steroid treatment and have shown clinical and radiographic stability for at least 14 days after definitive therapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 9-ING-41, gemcitabine, docetaxel, or other agents used in study.
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has had a previous (within 2 years) or has a current malignancy other than the target cancer with the exception of curatively treated local tumors including carcinoma in situ of the breast or cervix, basal or squamous cell carcinoma of the skin, or prostate cancer with Gleason Grade < 6 and prostate-specific antigen within normal range.
* Has any medical and/or social condition that, in the opinion of the investigator would preclude study participation.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate | Approximately 24 weeks
  To determine the Disease Control Rate (DCR = Complete Response [CR] + Partial Response [PR] + Stable Disease [SD] at 24 weeks) of 9-ING-41 in combination with gemcitabine and docetaxel in advanced sarcoma.

SECONDARY OUTCOMES:
Progression Free Survival | From start of protocol therapy, approximately 5 years
  To determine the activity of 9-ING-41 with chemotherapy by assessing progression free survival (PFS).

CONTACTS AND LOCATIONS:
Overall Officials: Bradley D DeNardo, MD, Principal Investigator — Brown University; Galina G Lagos, MD, Principal Investigator — Lifespan Cancer Institute
Locations (2):
- United States (2):
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Lifespan Cancer Insitute, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No